CLINICAL TRIAL: NCT02972151
Title: Clinical Promotion Research of Complex Treatment With TCM to Diagnosis and Treatment on Different Syndrome Types of Pelvic Inflammatory Disease Sequelae
Brief Title: Clinical Research of TCM on Pelvic Inflammatory Disease Sequelae
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 42501190
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Pelvic Inflammatory Disease
MeSH Terms: conditions — Pelvic Inflammatory Disease | interventions — Oral Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comprehensive treatment of TCM (Experimental): The intervention is Comprehensive treatment of TCM,which including Oral medicine ,tradition chinese medicine enema, external treatment.
  Interventions: Drug: Comprehensive treatment of TCM
- Expectant therapy (Active Comparator): Expectant treatment group patients were not treated during the observation period.
  （3 months after the start of the trial and 1 months after the end of the trial.）
  Interventions: Other: Expectant treatment

INTERVENTIONS:
Drug: Comprehensive treatment of TCM — Subjects were treated with comprehensive treatment of TCM including Oral medicine: 1 dose daily by our hospital pharmacy medicine room Decoction decoction, each agent 200ml, and the 2 ton service. 10 days for a course of treatment, continuous treatment of 3 courses; retention enema with traditional Chinese medicine oral drugs according to different types of concentrated decoction enema, each dose of medicine decocting 2 times, 2 days of external application of Chinese medicine: Chinese medicine enema; break into powder, into the bag, steam for 45 minutes, and so the temperature dropped to appropriate, will be installed a Chinese medicine bag used on patients with lower abdomen for 20 minutes. Above method, a course of treatment for 10 days, continuous treatment of 3 courses.
  Other Names: Oral medicine and TCM enema, external treatment
  Arms: Comprehensive treatment of TCM
Other: Expectant treatment — Expectant treatment group patients were not treated during the observation period.（3 months after the start of the trial and 1 months after the end of the trial.）From the point of view of medical ethics, the expectant treatment group of patients at the end of the observation period, given the treatment of traditional Chinese medicine treatment group.
  Other Names: Do not give any treatment
  Arms: Expectant therapy

SUMMARY:
The trial attempts to optimize, standardize and simplify the characteristic diagnosis and treatment program of the dominant diseases in our hospital-the sequelae of pelvic inflammatory disease, so as to make it suitable for clinical diagnosis and treatment in primary hospital.

DETAILED DESCRIPTION:
Sequelae of pelvic inflammatory disease (SPID) is a common cause of chronic pelvic pain, ectopic pregnancy and infertility, which seriously affects the physical and mental health of the patients, quality of life and family happiness. Western medicine for pelvic inflammatory disease sequelae is still lack of effective treatment methods, traditional Chinese medicine treatment of this disease has a unique advantage, with broad prospects for development..Standardized diagnosis and treatment scheme of this project on the one hand, improve and optimize the sequelae of pelvic inflammatory disease, including according to the dialectical treatment of herbal medicine combined with TCM (traditional Chinese medicine enema, external application of Chinese medicine intervention treatment); on the other hand, to observe the clinical curative effect and adverse reaction of traditional Chinese medicine comprehensive treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnostic criteria for the sequelae of pelvic inflammatory disease in Western medicine;
2. Patients conforming to the criteria of TCM syndrome differentiation;
3. Age 18--60 years old, married or sexual life;
4. In this study, the voluntary participation, and signed informed consent;

Exclusion Criteria:

1. Patients who do not meet the diagnostic criteria of Western medicine and traditional Chinese medicine dialectical typing standard;
2. Persons with acute pelvic inflammatory disease;
3. Related symptoms caused by diseasesGynecological tumor，specific vaginitis, acute cervicitis, pelvic congestion syndrome, endometriosis, adenomyosis, pelvic tuberculosis etc.
4. Pregnant and lactating women;
5. With severe primary disease, such as liver, kidney, heart, brain and hematopoietic system;
6. Allergic to a variety of drugs or known to be allergic to the composition of the use of traditional Chinese Medicine;
7. Patients taking part in other clinical trials;
8. Suspect or do have a history of alcohol, drug abuse or according to the judgment of the researcher,other lesions or circumstances that have reduced the likelihood of entering a group or the complexity of entering a group,such as frequent changes in the working environment, the living environment is not stable,etc.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
changes of The Symptom score | 3 months after treatment
  Patients are checked The Symptom score at 3 months after treatment.

SECONDARY OUTCOMES:
changes of The Hamilton Depression Scale (HAMD) (17 items) | 1 months after treatment, 2 months after treatment, 3 months after treatment and 1 months after drug withdrawal.
changes of The Sign score sheet | 1 months after treatment, 2 months after treatment, 3 months after treatment and 1 months after drug withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: lianwei xu, Doctor, Principal Investigator — Shanghai Longhua Hospital
Locations (1):
- Shanghai Longhua Hosptial, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No